CLINICAL TRIAL: NCT06583772
Title: Validity and Reliability of the BeCureTM Virtual Reality-Based 9-Hole Peg Test in Stroke Patients
Brief Title: Validity and Reliability of the Virtual Reality-Based 9-Hole Peg Test in Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Haydar Gok, Professor Doctor, Ankara University
Other Study IDs: I02-56-23
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: stroke; Virtual reality; Nine-hole peg test
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Post-stroke patients
  Interventions: Diagnostic Test: VR-based 9-hole peg test

INTERVENTIONS:
Diagnostic Test: VR-based 9-hole peg test — The volunteers will first undergo a physical 9-hole peg test. After the physical test is completed, the VR-based 9-hole peg test will be performed.

SUMMARY:
The goal of this observational study is to demonstrate diagnostic value of a VR-based 9-hole peg test (9HPT) for the evaluation of manual dexterity in stroke patients.

The main questions it aims to answer are:

* Is the VR-based 9HPT a reliable and valid diagnostic tool to evaluate manual dexterity in stroke patients when compared to the physical version of it.
* Does the VR-based 9HPT differ between the dominant and non-dominant hand in healthy individuals?

DETAILED DESCRIPTION:
The 9-hole peg test (9HPT) is a method used to assess finger dexterity in patients with various neurological diseases, including stroke, Parkinson's disease, and cerebral palsy. Additionally, this test evaluates strength, visual attention, depth perception, sensory perception, and motor coordination.

The psychometric properties of the 9HPT were evaluated in healthy normal subjects and stroke patients in various studies. The results of these suggest that the 9HPT may be a reliable, valid and responsive measure in patients with stroke. Although the test is relatively straightforward to administer, it does have a number of disadvantages. The patient may knock over the test tools, take more than one peg at a time, use both hands, start to remove the pegs back before filling all the holes, or drop the pegs on the floor. Furthermore, errors in time measurement may occur due to the tester performance. The latest developments in technology have led to the creation of electronic and virtual reality (VR) based versions of the 9HPT. These new versions have eliminated the disadvantages of the original test, allow for the storage of measurement results, and provide a way to track the treatment process both in the hospital and remotely. However, studies on the validity and reliability of these tests in individuals with neurological diseases remain limited. The aim of this study is therefore to demonstrate the validity and reliability of a VR-based 9HPT for the evaluation of manual dexterity in stroke patients. The secondary aims were to determine the normative values of the test in healthy individuals and to reveal whether there is a difference between the dominant and non-dominant hand.

The study is a cross-sectional observational trial. Post-stroke patients who applied to the Ankara University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation will be included in the study. Socio-demographic data such as gender, age, education level, occupation, background, duration of stroke, type of lesion, and history of comorbidities will be recorded. All patients will be evaluated at the beginning and after 7 days. The state of consciousness, orientation and cooperation will be evaluated on the physical examination and the patients will be given a Mini Mental Test. Participants who score 22 points or more on this assessment will be included in this study. Brunnstrom motor staging will be performed for motor assessment of stroke patients. The Modified Ashworth Scale will be used to assess spasticity. Accordingly, participants with spasticity grade 3 and above in the upper extremity will be excluded from the study. The participants will first undergo a physical 9HPT. After the physical test is completed, a VR-based 9HPT will be performed. A laptop computer, motion controller, and BecureTM software will be used for this purpose. Through a motion sensor (Leap Motion Controller) positioned on the table and not touching the participant, the upper extremity and hand movements will be reflected on the computer screen. During the test, participants will first practice 2 times and then be tested. The test will be repeated 3 times and the average value will be recorded in seconds. The test will be repeated in the same way after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a stroke diagnosis according to the WHO definition
* Upper extremity in stage 3 and above according to Brunnstrom motor staging
* To be cognitively competent (score of 22 or above on the Mini Mental Test)
* Balance of sitting
* The patient or his/her relatives have completed the informed voluntary consent form

Exclusion Criteria:

* Presence of severe aphasia
* Presence of cognitive impairment or psychiatric disorders
* Detection of a neglect phenomenon
* Presence of hemianopsia
* Spasticity in the affected arm, 3 or more according to Modified Ashworth Scale

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-stroke patients consecutively admitted to Ankara University Faculty of Medicine, Department of Physical Medicine and Rehabilitation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability of the VR-based 9-hole peg test | Baseline and 7 days
  Scoring is based on the time taken to complete the VR based 9-hole peg test activity, recorded in seconds. The volunteers will first undergo a physical 9-hole peg test. After the physical test is completed, the VR-based 9-hole peg test will be performed. In this application, patients will first practice 2 times and then be tested. The test will be repeated 3 times and the average value will be recorded in seconds. The test will be repeated in the same way after 7 days. To determine the reliability of the test, an intra-class correlation coefficient-ICC will be calculated.

SECONDARY OUTCOMES:
Internal consistency of the VR-based 9-hole test | Baseline
  Scoring is based on the time taken to complete the VR based 9-hole peg test activity, recorded in seconds. The volunteers will first undergo a physical 9-hole peg test. After the physical test is completed, the VR-based 9-hole peg test will be performed. In this application, patients will first practice 2 times and then be tested. The test will be repeated 3 times and the average value will be recorded in seconds. To determine the internal consistency of the test, Cronbach's alpha coefficient will be calculated.
Construct validity of the VR-based 9-hole test | Baseline
  Scoring is based on the time taken to complete the VR based 9-hole peg test activity, recorded in seconds. The volunteers will first undergo a physical 9-hole peg test. After the physical test is completed, the VR-based 9-hole peg test will be performed. The criterion validity of the test will be calculated by its agreement with the physical 9-hole peg test (Spearman's rank correlation).
To determine the normative values of the virtual reality-based 9-hole peg test in healthy individuals and to reveal whether there is a difference between dominant and non-dominant hand. | Baseline
  In age- and gender-matched healthy volunteers, the VR-based 9-hole peg test test will be performed on both the dominant and non-dominant hand. Scoring is based on the time taken to complete the VR based 9-hole peg test activity, recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Gok, Professor, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)